CLINICAL TRIAL: NCT05151978
Title: Transcranial Doppler as an Early Predictor of Neurological Outcome in Mild and Moderate Traumatic Brain Injury
Brief Title: Transcranial Doppler in Mild and Moderate Traumatic Brain Injury (TBI)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mai Kamal, Tanta elnady street elgharbia, Tanta University
Other Study IDs: 33574/12/19
Record Dates: First submitted 2021-11-26; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Trauma, Brain
Keywords: Trans , cranial, TBI
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- (glasgow coma scale) 9 _15: No Secondary Neurological deterioration
  Interventions: Diagnostic Test: Transcranial Doppler
- (glasgow coma scale) 9_15: Secondary Neurological deterioration
  Interventions: Diagnostic Test: Transcranial Doppler

INTERVENTIONS:
Diagnostic Test: Transcranial Doppler — Transcranial Doppler on middle cerebral arteries
  Other Names: CT of the brain

SUMMARY:
Utility of transcranial Doppler as an Early Predictor of Neurological deterioration in Mild and Moderate Traumatic Brain Injury

DETAILED DESCRIPTION:
Transcranial Doppler done to TBI patients on admission and follow up was done and Secondary Neurological deterioration was documented

ELIGIBILITY:
Inclusion Criteria:

* patient with traumatic brain injury and glasgow coma scale 9_15

Exclusion Criteria:

Unstable or patient on Mechanical ventilation, Sever brain injury , patient receive anticoagulant

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient with TBI
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-02-22 (Estimated)

PRIMARY OUTCOMES:
Secondary Neurological deterioration | 7 days
  Decrease in glasgow coma scale and /or deterioration need to surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Goneim, Study Chair — Head of faculty of medicine
Locations (1):
- Faculty of Medicine, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data of transcranial Doppler of middle cerebral arteries and the Neurological outcome
Supporting Information: Study Protocol, SAP
Time Frame: From October 2021 till December 2022
Access Criteria: All data collected after statistical analysis

REFERENCES:
- See also: https://pubmed.ncbi.nlm.nih.gov/31497078/ — https://pubmed.ncbi.nlm.nih.gov/31497078/

DOCUMENTS (1):
  • Study Protocol (2021-01-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT05151978/Prot_000.pdf